CLINICAL TRIAL: NCT06780657
Title: The Effect of Hypopressive Exercise on Overactive Bladder Syndrome and Quality of Life
Brief Title: Overactive Bladder Syndrome and Hypopressive Exercise
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sevgi Özkan, Dean of Health Sciences, Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-60116787-020-548394
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Overactive Bladder Syndrome
Keywords: Overactive Bladder Syndrome; Overactive Bladder; Hypopressive Exercise; Quality of Life
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Women who meet the inclusion criteria will be distributed to the experimental and control groups in a randomized controlled manner.
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive an online hypopressive exercise training program for 8 weeks.
  Interventions: Behavioral: Online hypopressive exercise training program
- Control Group (No Intervention): No special intervention.

INTERVENTIONS:
Behavioral: Online hypopressive exercise training program — The hypopressive exercises were based on recommendations from the literature and consultation with an expert in the field. Each session will be held twice a week for 20-25 minutes. Participants will perform each exercise 10 times during these sessions.
  Arms: Experimental Group

SUMMARY:
Overactive Bladder Syndrome (OAB) is a condition characterized by a sudden and urgent need to urinate, with or without urge incontinence, accompanied by increased urinary frequency. This syndrome significantly impacts individuals' social and economic lives, psychological well-being, work productivity, daily activities, and overall quality of life.

The Abdominal Hypopressive Technique (AHT) was suggested by Caufriez for the treatment of pelvic floor disorders in women. It has been utilized in the treatment of pelvic floor dysfunctions, such as Urinary Incontinence (UI), particularly in postpartum women.

A review of the existing literature reveals a lack of studies examining the relationship between overactive bladder syndrome and hypopressive exercises. Current research predominantly focuses on the effects of hypopressive exercises on pelvic organ prolapse, pelvic floor muscle tone, urinary incontinence, and stress urinary incontinence. Although AHT was initially developed for the treatment of pelvic floor disorders, it is now recommended for all women, regardless of the presence of UI. However, studies on AHT remain limited, which poses challenges for its broader scientific application. This highlights the need for robust scientific studies to strengthen the evidence base. The present study aims to evaluate the impact of an online hypopressive exercise training program on overactive bladder syndrome symptoms and quality of life. The main questions it aims to answer are:

* Does online hypopressive exercise training effectively reduce the symptoms of overactive bladder syndrome?
* Does online hypopressive exercise training effective in improving the quality of life among women with overactive bladder syndrome?

DETAILED DESCRIPTION:
The study was designed as a prospective, single-blind, randomized controlled experimental trial with a pretest-posttest control group design. The study sample consisted of women diagnosed with Overactive Bladder Syndrome (OAB) who applied to the Urology Outpatient Clinic of Pamukkale University Hospital and those reached via social media (scoring above 11 on the Overactive Bladder Screening Form [OAB-V8]). Eligibility was determined using a personal information form, the Overactive Bladder Screening Form (OAB-V8), and the Overactive Bladder Quality of Life Questionnaire (OAB-q).

The contact information of women in the experimental and control groups was collected, and data were gathered through Google Forms, with online communication established via messaging. To reach participants through social media, a poster was prepared, and the online hypopressive exercise training program was announced. All participants were verbally informed about the study via the details provided in the informed consent form, and verbal consent was obtained. Additionally, an explanation was provided in the initial section of the data form, and women who agreed to participate clicked "I voluntarily agree to participate in the study" to access the form.

The sample size was calculated using the G Power 3.1.9.4 software with an a priori power analysis. Considering a power of 80% and a 10% excess for potential sample loss, a minimum of 56 participants per group was determined. Simple randomization was used for this study.

The hypopressive exercises used in this study were determined based on recommendations from the literature and consultation with an expert in the field. Participants in the experimental group were asked to complete the relevant scales via Google Forms before starting the online hypopressive exercise training (pretest). They were then instructed to perform the exercises twice a week for 20-25 minutes over eight weeks, repeating each exercise 10 times per session by the end of the program. They were also asked to mark their progress on an 8-week exercise diary. After the eight weeks, they were requested to complete the same scales via Google Forms again (posttest).

Participants in the control group were asked to maintain their usual physical activities and continue with their normal daily lives. At the end of the eight weeks, they were also requested to complete the same scales via Google Forms (posttest).

The outcomes were measured at the start of the intervention and after eight weeks. Data were collected using the personal information form, the Overactive Bladder Screening Form (OAB-V8), and the Overactive Bladder Quality of Life Questionnaire (OAB-q).

ELIGIBILITY:
Inclusion Criteria:

* No contraindications to performing hypopressive exercises,
* Voluntary participation in the study,
* Being between 18 and 65 years of age,
* Having access to the internet,
* Ability to speak and understand Turkish.

Exclusion Criteria:

* Individuals with lower back pain,
* Those with uncontrolled hypertension,
* Individuals with hiatal hernia,
* Those with a history of inguinal hernia,
* Pregnant individuals,
* Those diagnosed with COPD,
* Individuals with neuromuscular disorders,
* Those who have undergone abdominal or pelvic surgery,
* Prior experience with hypopressive exercises.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 112 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Overactive Bladder Evaluation Form (OAB-V8) | At the end of 8 weeks
  It is a scale consisting of 8 questions, each with 6 options on a Likert type scale (Not at all-0, very little-1, a little-2, a lot-3, a lot-4, a lot-5) to question the presence of Overactive Bladder Syndrome. The total score is between 0-40. Accordingly, those with a total score of >11 are classified as Overactive Bladder Syndrome patients.

SECONDARY OUTCOMES:
Overactive Bladder Quality of Life Scale (OAB-q) | At the end of 8 weeks
  OAB-q is a quality of life scale consisting of 33 questions that evaluate symptom severity and health-related quality of life in patients with overactive bladder syndrome (OAMS). Each consists of 6 Likert-type options (Never-1, Rarely-2, Sometimes-3, Somewhat often-4, Often-5, Always-6) and 4 subcategories (coping, anxiety, sleep and social relationships). It has a score assessment ranging from 0 to 100. An increase in symptom discomfort indicates an increase in symptom severity, while an increase in quality of life score is a good sign.

OTHER OUTCOMES:
Personal information form | Baseline
  The form was designed by researchers to learn the sociodemographic characteristics of women and their pregnancy status (nulliparous, multiparous), number of pregnancies, number of births, type of birth (vaginal, cesarean, vaginal-cesarean), use of cigarettes, alcohol, acidic/carbonated drinks, coffee-nescafe, herbal tea, spicy foods, artificial sweeteners, depression status and physical activity status.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Resende APM, Bernardes BT, Stupp L, Oliveira E, Castro RA, Girao MJBC, Sartori MGF. Pelvic floor muscle training is better than hypopressive exercises in pelvic organ prolapse treatment: An assessor-blinded randomized controlled trial. Neurourol Urodyn. 2019 Jan;38(1):171-179. doi: 10.1002/nau.23819. Epub 2018 Oct 12. PMID 30311680
- [Background] Navarro Brazalez B, Sanchez Sanchez B, Prieto Gomez V, De La Villa Polo P, McLean L, Torres Lacomba M. Pelvic floor and abdominal muscle responses during hypopressive exercises in women with pelvic floor dysfunction. Neurourol Urodyn. 2020 Feb;39(2):793-803. doi: 10.1002/nau.24284. Epub 2020 Jan 27. PMID 31985114
- [Background] Soriano L, Gonzalez-Millan C, Alvarez Saez MM, Curbelo R, Carmona L. Effect of an abdominal hypopressive technique programme on pelvic floor muscle tone and urinary incontinence in women: a randomised crossover trial. Physiotherapy. 2020 Sep;108:37-44. doi: 10.1016/j.physio.2020.02.004. Epub 2020 Feb 19. PMID 32707289
- [Background] Molina-Torres G, Moreno-Munoz M, Rebullido TR, Castellote-Caballero Y, Bergamin M, Gobbo S, Hita-Contreras F, Cruz-Diaz D. The effects of an 8-week hypopressive exercise training program on urinary incontinence and pelvic floor muscle activation: A randomized controlled trial. Neurourol Urodyn. 2023 Feb;42(2):500-509. doi: 10.1002/nau.25110. Epub 2022 Dec 8. PMID 36482844
- [Background] Jose-Vaz LA, Andrade CL, Cardoso LC, Bernardes BT, Pereira-Baldon VS, Resende APM. Can abdominal hypropressive technique improve stress urinary incontinence? an assessor-blinded randomized controlled trial. Neurourol Urodyn. 2020 Nov;39(8):2314-2321. doi: 10.1002/nau.24489. Epub 2020 Aug 19. PMID 32813928
- [Background] Ithamar L, de Moura Filho AG, Benedetti Rodrigues MA, Duque Cortez KC, Machado VG, de Paiva Lima CRO, Moretti E, Lemos A. Abdominal and pelvic floor electromyographic analysis during abdominal hypopressive gymnastics. J Bodyw Mov Ther. 2018 Jan;22(1):159-165. doi: 10.1016/j.jbmt.2017.06.011. Epub 2017 Jun 21. PMID 29332741